CLINICAL TRIAL: NCT04000880
Title: Adapting MultiPLe Behavior Interventions That eFfectively Improve (AMPLIFI) Cancer Survivor Health
Brief Title: Adapting Multiple Behavior Interventions That Effectively Improve Cancer Survivor Health Cancer Survivor Health
Acronym: AMPLIFY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Tennessee (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wendy Demark-Wahnefried, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB-300002068; 1P01CA229997 (NIH)
Record Dates: First submitted 2019-06-21; First posted 2019-06-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Colorectal Cancer; Endometrial Cancer; Kidney Cancer; Multiple Myeloma; Ovary Cancer; Prostate Cancer; Thyroid Cancer; Non-Hodgkin Lymphoma
Keywords: Cancer survivor; Lifestyle behaviors; Web-based intervention; Diet; Exercise; Weight Control; Physical Activity; Distance Medicine; Rural; Older; Minority; African American
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Kidney Neoplasms; Multiple Myeloma; Ovarian Neoplasms; Prostatic Neoplasms; Thyroid Neoplasms; Lymphoma, Non-Hodgkin; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will participate in one of three arms:
  1. Diet followed by Exercise intervention
  2. Exercise followed by Diet intervention
  3. Combined Diet and Exercise intervention
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Single blinded trial in which the study participant and select individuals in the research team (i.e., interventionists) will be aware of randomization status, but the assessors and investigators will not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Project 1: Diet-Exercise (Experimental): Participants will receive and participate in web-based sessions that focus on diet for 6 months, followed by exercise for another 6 months. Participants will be encouraged to track their diet and weight for the first 6 months and to log their data in the intervention website, during the second 6 months they will be asked to log their physical activity data (minutes and step counts). Tailored feedback and goal recommendations will be provided through the website. Participants will also receive access to resources for relevant behavioral topics. All participants will be invited to participate in the secret Facebook group for the project (though participation is optional).
  Interventions: Behavioral: Adapting MultiPLe Behavior Interventions That eFfectively Improve (AMPLIFI) Cancer Survivor Health; Other: Combined Diet and Exercise
- Project 2: Exercise-Diet (Experimental): Participants will receive and participate in web-based sessions that focus on diet for 6 months, followed by exercise for another 6 months. Participants will be encouraged to track their diet and weight for the first 6 months and to log their data in the intervention website, during the second 6 months they will be asked to log their physical activity data (minutes and step counts). Tailored feedback and goal recommendations will be provided through the website. Participants will also receive access to resources for relevant behavioral topics. All participants will be invited to participate in the secret Facebook group for the project (though participation is optional).
  Interventions: Behavioral: Adapting MultiPLe Behavior Interventions That eFfectively Improve (AMPLIFI) Cancer Survivor Health; Other: Combined Diet and Exercise
- Project 3: Combined Diet and Exercise (Experimental): Participants will receive the diet and exercise content simultaneously in combined web-based sessions. Participants will receive and participate in web-based sessions that focus on diet and exercise for 12 months. Participants will be encouraged to track their diet, weight and physical activity data (minutes and step counts). Tailored feedback and goal recommendations will be provided through the website. Participants will also receive access to resources for relevant behavioral topics. All participants will be invited to participate in the secret Facebook group for the project (though participation is optional).
  Interventions: Behavioral: Adapting MultiPLe Behavior Interventions That eFfectively Improve (AMPLIFI) Cancer Survivor Health; Other: Diet-Exercise; Other: Exercise-Diet

INTERVENTIONS:
Behavioral: Adapting MultiPLe Behavior Interventions That eFfectively Improve (AMPLIFI) Cancer Survivor Health — AMPLIFI will provide participants with a secure website where they receive and participate in educational sessions tailored to their assigned topics for the intervention arm. The website will provide a resource library for static documents, tips of the day, tracking of health behaviors, and goal-setting.
  Other Names: AiM, Plan and act on LIFestYles: AMPLIFY Survivor Health
Other: Diet-Exercise — Diet-Exercise
  Arms: Project 3: Combined Diet and Exercise
Other: Exercise-Diet — Exercise-Diet
  Arms: Project 3: Combined Diet and Exercise
Other: Combined Diet and Exercise — Combined Diet and Exercise
  Arms: Project 1: Diet-Exercise; Project 2: Exercise-Diet

SUMMARY:
This research study will test the efficacy of interactive, web-based interventions that improve diet, physical activity and weight management changes among early stage survivors of breast, prostate, colorectal, endometrial, renal, thyroid, and ovarian cancers, as well as multiple myeloma and non-Hodgkin Lymphoma. Overarching outcomes also include physical function and performance, muscle mass, quality of life, and health utilities.

DETAILED DESCRIPTION:
For this web-based behavioral intervention trial aimed at improving lifestyle behaviors of individuals at higher risk for cancer, other comorbidities and functional decline, 652 cancer survivors (a large proportion of whom will be age 65 or over, rural, and of minority status) will be enrolled and randomly assigned to one of the following study arms: 1) A diet and exercise intervention which would begin immediately, with the first 6 months focused on promoting healthful changes in diet consistent with the American Institute for Cancer Research Guidelines and designed to invoke an average weight loss of one pound per week, and the second 6 months focused on increasing physical activity. The 163 cancer survivors assigned to this arm would be evaluated at baseline, 6-, 12- and 18-months; 2) An exercise and diet intervention which would begin immediately, with the first 6 months focused on increasing physical activity, and the second 6 months focused on promoting healthful changes in diet consistent with the American Institute for Cancer Research Guidelines and designed to invoke an average weight loss of one pound per week. The 163 cancer survivors assigned to this arm would be evaluated at baseline, 6-, 12- and 18-months; and 3) A 12-month combined diet and exercise intervention focused on promoting healthful changes in diet consistent with the American Institute for Cancer Research Guidelines and designed to invoke an average weight loss of one pound per week, while at the same time promoting physical activity. The 326 cancer survivors assigned to this arm will be evaluated at baseline, 6-, 12-, and 18-months. Weight status, waist circumference, body composition, diet quality, physical activity, physical performance, quality of life, comorbidity, and health utilities will be measured at baseline and each follow-up time point, as will mediators of behavior change, e.g., social support, self-efficacy and barriers. Additionally, dried blood spots obtained from fingersticks will be analyzed for cytokines (IL-6 and hsCRP) and biomarkers of gluco- and lipid regulation, i.e., glucose, and blood lipids (TG) and insulin.

It is hypothesized that cancer survivors assigned to all three of these study arms will experience significant improvements in weight status, body composition, diet quality, physical activity, physical performance, and quality of life. These improvements also will translate into lower health utility scores and prove cost effective. It also is anticipated that analyses will uncover significant mediators, such as self-efficacy, and moderators, such as level of educational attainment associated with program efficacy. Finally, we hypothesize that while all study arms will experience significant benefit, the sequenced arm participants (arms 1 and 2) will have significantly greater odds of achieving improved diet quality, weight loss, and moderate intensity aerobic physical activity of at least 150 minutes a week as measured by accelerometer) post-intervention than survivors randomized to the simultaneous arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Resident of the continental United States
* Diagnosed with multiple myeloma, non-Hodgkin lymphoma, or localized kidney or ovarian cancer; or [localized (includes in situ) through regional] breast, colorectum, endometrium, thyroid, or prostate cancer.
* Completed primary treatment (surgery, radiation or chemotherapy). Active surveillance among men with prostate cancer or women with ductal carcinoma in situ is acceptable.
* Completion of the 8th grade of school. Able to read and write English.
* Normal blood pressure or those with high blood pressure for whom physician permission was granted.
* Community dwelling.
* Reside in an area that receives wireless coverage.
* Have an active email address or be willing to have one created for the study.
* Current body mass index of greater than or equal to 25 kg/m2, but less than 50 kg/m2.
* Current physical activity level is less than 150 minutes of moderate-to-vigorous exercise per week.

Exclusion Criteria:

* Participation in another diet and exercise program.
* Evidence of progressive cancer of the eligible types.
* Recurrence of the eligible cancer types (exceptions are biochemical recurrence of prostate cancer).
* A physician has provided instruction to limit current physical activity.
* Pre-existing medical conditions that preclude adherence to an unsupervised weight loss intervention (e.g., pregnancy, severe orthopedic conditions, impending hip or knee replacement (within 6 months), end-stage renal disease, paralysis, dementia, blindness, unstable angina, untreated stage 3 hypertension, or recent history of heart attack, congestive heart failure or pulmonary conditions that required oxygen or hospitalization within 6 months).
* Second primary cancers, with the exception of non-melanoma skin cancer, or if the initial and second cancers are both deemed eligible cancers.
* Reside in a skilled nursing or assisted living facility.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in dietary quality and intake (Patient reported outcome). | Baseline
  Participants will complete two dietary recalls (one weekday and one weekend day)
Change in dietary quality and intake (Patient reported outcome). | 6 months
  Participants will complete two dietary recalls (one weekday and one weekend day)
Change in dietary quality and intake (Patient reported outcome). | 12 months
  Participants will complete two dietary recalls (one weekday and one weekend day)
Change in dietary quality and intake (Patient reported outcome). | 18 months
  Participants will complete two dietary recalls (one weekday and one weekend day)
Change in dietary quality and intake (Patient reported outcome). | 24 months
  Participants will complete two dietary recalls (one weekday and one weekend day)
Change in body weight | Baseline
  Participant body weight will be measured during an in-person or remote (Zoom) visit
Change in body weight | 6 months
  Participant body weight will be measured during an in-person or remote (Zoom) visit
Change in body weight | 12 months
  Participant body weight will be measured during an in-person or remote (Zoom) visit
Change in body weight | 18 months
  Participant body weight will be measured during an in-person or remote (Zoom) visit
Change in body weight | 24 months
  Participant body weight will be measured during an in-person or remote (Zoom) visit
Change in physical activity and sleep (Measured by actigraphy) | Baseline
  Physical activity and sleep will be measured objectively via blank screen accelerometers which are small devices (1x2 inches) that will be worn at the waist during waking hours and switched to a wrist band during sleep for a 7-day period at each assessment point.
Change in physical activity and sleep (Measured by actigraphy) | 6 months
  Physical activity and sleep will be measured objectively via blank screen accelerometers which are small devices (1x2 inches) that will be worn at the waist during waking hours and switched to a wrist band during sleep for a 7-day period at each assessment point.
Change in physical activity and sleep (Measured by actigraphy) | 12 months
  Physical activity and sleep will be measured objectively via blank screen accelerometers which are small devices (1x2 inches) that will be worn at the waist during waking hours and switched to a wrist band during sleep for a 7-day period at each assessment point.
Change in physical activity and sleep (Measured by actigraphy) | 18 months
  Physical activity and sleep will be measured objectively via blank screen accelerometers which are small devices (1x2 inches) that will be worn at the waist during waking hours and switched to a wrist band during sleep for a 7-day period at each assessment point.
Change in physical activity and sleep (Measured by actigraphy) | 24 months
  Physical activity and sleep will be measured objectively via blank screen accelerometers which are small devices (1x2 inches) that will be worn at the waist during waking hours and switched to a wrist band during sleep for a 7-day period at each assessment point.

SECONDARY OUTCOMES:
Change in waist circumference | Baseline
  Waist circumference will be measured using unmarked tapes at the level of the umbilicus during the in-person or remote assessments.
Change in waist circumference | 6 months
  Waist circumference will be measured using an unmarked tape at the level of the umbilicus during the in-person or remote assessments.
Change in waist circumference | 12 months
  Waist circumference will be measured using an unmarked tape at the level of the umbilicus during in-person or remote assessments.
Change in waist circumference | 18 months
  Waist circumference will be measured using an marked tape at the level of the umbilicus during the in-person or remote assessments.
Change in waist circumference | 24 months
  Waist circumference will be measured using an unmarked tape at the level of the umbilicus during the in-person or remote assessments.
Change in muscle mass (Measured by the D3 creatine dilution method) | Baseline
  To assess muscle mass, participants will take a capsule containing deuterium-labelled creatine [creatine is a substance commonly found in protein-containing foods and deuterium is a naturally-occurring element], the administration of which is proven as safe with several studies conducted in humans across the lifespan from pre-term infants to elders and will use a urine test strip 3 days later on their 2nd void of the day
Change in muscle mass (Measured by the D3 creatine dilution method) | 6 months
  To assess muscle mass, participants will take a capsule containing deuterium-labelled creatine [creatine is a substance commonly found in protein-containing foods and deuterium is a naturally-occurring element], the administration of which is proven as safe with several studies conducted in humans across the lifespan from pre-term infants to elders and will use a urine test strip 3 days later on their 2nd void of the day
Change in muscle mass (Measured by the D3 creatine dilution method) | 12 months
  To assess muscle mass, participants will take a capsule containing deuterium-labelled creatine [creatine is a substance commonly found in protein-containing foods and deuterium is a naturally-occurring element], the administration of which is proven as safe with several studies conducted in humans across the lifespan from pre-term infants to elders and will use a urine test strip 3 days later on their 2nd void of the day
Change in muscle mass (Measured by the D3 creatine dilution method) | 18 months
  To assess muscle mass, participants will take a capsule containing deuterium-labelled creatine [creatine is a substance commonly found in protein-containing foods and deuterium is a naturally-occurring element], the administration of which is proven as safe with several studies conducted in humans across the lifespan from pre-term infants to elders and will use a urine test strip 3 days later on their 2nd void of the day
Change in muscle mass (Measured by the D3 creatine dilution method) | 24 months
  To assess muscle mass, participants will take a capsule containing deuterium-labelled creatine [creatine is a substance commonly found in protein-containing foods and deuterium is a naturally-occurring element], the administration of which is proven as safe with several studies conducted in humans across the lifespan from pre-term infants to elders and will use a urine test strip 3 days later on their 2nd void of the day
Change in physical performance | Baseline
  Participants will complete the Senior Fitness Battery during the in-person or remote assessments, which includes chair stands, 3m walk, 8' up and go, balance testing (side-by-side, semi-tandem and tandem stances), reaching (stretching exercises of the arms and legs, and the 2-minute step test.
Change in physical performance | 6 Months
  Participants will complete the Senior Fitness Battery during the in-person or remote assessments, which includes chair stands, 3m walk, 8' up and go, balance testing (side-by-side, semi-tandem and tandem stances), reaching (stretching exercises of the arms and legs, and the 2-minute step test.
Change in physical performance | 12 months
  Participants will complete the Senior Fitness Battery during the in-person or remote assessments, which includes chair stands, 3m walk, 8' up and go, balance testing (side-by-side, semi-tandem and tandem stances), reaching (stretching exercises of the arms and legs, and the 2-minute step test.
Change in physical performance | 18 months
  Participants will complete the Senior Fitness Battery during the in-person or remote assessments, which includes chair stands, 3m walk, 8' up and go, balance testing (side-by-side, semi-tandem and tandem stances), reaching (stretching exercises of the arms and legs, and the 2-minute step test.
Change in physical performance | 24 months
  Participants will complete the Senior Fitness Battery during the in-person or remote assessments, which includes chair stands, 3m walk, 8' up and go, balance testing (side-by-side, semi-tandem and tandem stances), reaching (stretching exercises of the arms and legs, and the 2-minute step test.
Change in physical activity (Patient reported outcome) | Baseline
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 3 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 6 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 9 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 12 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 15 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 18 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 21 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in physical activity (Patient reported outcome) | 24 months
  Physical activity will be measured via validated questionnaires (e.g., the Godin Leisure Time Physical Activity and the Global Physical Activity Questionnaires).
Change in quality of life (Patient reported outcome) | Baseline
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 3 Months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 6 Months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 9 Months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 12 months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 15 months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 18 months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 21 months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in quality of life (Patient reported outcome) | 24 months
  Participants will complete questionnaires (PROMIS Cancer-Related Item Bank and Short Form 12) to self-report quality of life.
Change in healthcare utilization (Patient reported outcome) | Baseline
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 3 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 6 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 9 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 12 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 15 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 18 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 21 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.
Change in healthcare utilization (Patient reported outcome) | 24 months
  Participants will complete a healthcare utilization survey to capture physician and emergency room visits, and hospitalizations.

OTHER OUTCOMES:
Change in Levels of Stress (Patient reported outcome) | baseline
  Participants will complete the 14-item Perceived Stress Scale
Change in Levels of Stress (Patient reported outcome) | 6 months
  Participants will complete the 14-item Perceived Stress Scale
Change in Levels of Stress (Patient reported outcome) | 12 months
  Participants will complete the 14-item Perceived Stress Scale
Change in Levels of Stress (Patient reported outcome) | 18 months
  Participants will complete the 14-item Perceived Stress Scale
Change in Levels of Stress (Patient reported outcome) | 24 months
  Participants will complete the 14-item Perceived Stress Scale
Change in CIrculating Biomarkers | baseline
  Fingersticks done after a 12-hour fast will collect 5 blood spots which will be dried (DBS). DBS eluents will be batch-tested against known standards for insulin, glucose, leptin, adiponectin, high density lipoprotein and total cholesterol, tryglycerides, interleukin-6, c-reactive protein and tumor necrosis factor alpha
Change in CIrculating Biomarkers | 6 months
  Fingersticks done after a 12-hour fast will collect 5 blood spots which will be dried (DBS). DBS eluents will be batch-tested against known standards for insulin, glucose, leptin, adiponectin, high density lipoprotein and total cholesterol, tryglycerides, interleukin-6, c-reactive protein and tumor necrosis factor alpha
Change in CIrculating Biomarkers | 12 months
  Fingersticks done after a 12-hour fast will collect 5 blood spots which will be dried (DBS). DBS eluents will be batch-tested against known standards for insulin, glucose, leptin, adiponectin, high density lipoprotein and total cholesterol, tryglycerides, interleukin-6, c-reactive protein and tumor necrosis factor alpha
Change in CIrculating Biomarkers | 18 months
  Fingersticks done after a 12-hour fast will collect 5 blood spots which will be dried (DBS). DBS eluents will be batch-tested against known standards for insulin, glucose, leptin, adiponectin, high density lipoprotein and total cholesterol, tryglycerides, interleukin-6, c-reactive protein and tumor necrosis factor alpha
Change in CIrculating Biomarkers | 24 months
  Fingersticks done after a 12-hour fast will collect 5 blood spots which will be dried (DBS). DBS eluents will be batch-tested against known standards for insulin, glucose, leptin, adiponectin, high density lipoprotein and total cholesterol, tryglycerides, interleukin-6, c-reactive protein and tumor necrosis factor alpha
Change in Comorbidity and Symptoms (Patient reported outcome) | baseline
  The 43-item Older Americans Resources & Services (OARS) Questionnaire will be administered
Change in Comorbidity and Symptoms (Patient reported outcome) | 6 months
  The 43-item Older Americans Resources & Services (OARS) Questionnaire will be administered
Change in Comorbidity and Symptoms (Patient reported outcome) | 12 months
  The 43-item Older Americans Resources & Services (OARS) Questionnaire will be administered
Change in Comorbidity and Symptoms (Patient reported outcome) | 18 months
  The 43-item Older Americans Resources & Services (OARS) Questionnaire will be administered
Change in Comorbidity and Symptoms (Patient reported outcome) | 24 months
  The 43-item Older Americans Resources & Services (OARS) Questionnaire will be administered
Social Support, self-efficacy and barriers for adhering to a caloric restricted diet or increased PA (Patient Reported Outcomes) | baseline
  Validated items from Sallis et al, Clark, et al, Rogers, et al, McAiley, et al
Social Support, self-efficacy and barriers for adhering to a caloric restricted diet or increased PA (Patient Reported Outcomes) | 6 months
  Validated items from Sallis et al, Clark, et al, Rogers, et al, McAiley, et al
Social Support, self-efficacy and barriers for adhering to a caloric restricted diet or increased PA (Patient Reported Outcomes) | 12 months
  Validated items from Sallis et al, Clark, et al, Rogers, et al, McAiley, et al
Social Support, self-efficacy and barriers for adhering to a caloric restricted diet or increased PA (Patient Reported Outcomes) | 18 months
  Validated items from Sallis et al, Clark, et al, Rogers, et al, McAiley, et al
Social Support, self-efficacy and barriers for adhering to a caloric restricted diet or increased PA (Patient Reported Outcomes) | 24 months
  Validated items from Sallis et al, Clark, et al, Rogers, et al, McAiley, et al
Quality of Life, EQ-5D-5L | baseline
  comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Quality of Life, EQ-5D-5L | 6 months
  comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Quality of Life, EQ-5D-5L | 18 months
  comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Quality of Life, EQ-5D-5L | 24 months
  comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Health literacy and Ehealth literacy scales (eHEALS) | baseline
  The eHealth Literacy Scale measures (1) to assess consumers' perceived skills at using information technology for health and (2) to aid in determining the fit between eHealth programs and consumers. Norman, 2006
Health literacy and Ehealth literacy scales (eHEALS) | 6 months
  The eHealth Literacy Scale measures (1) to assess consumers' perceived skills at using information technology for health and (2) to aid in determining the fit between eHealth programs and consumers. Norman, 2006
Health literacy and Ehealth literacy scales (eHEALS) | 12 months
  The eHealth Literacy Scale measures (1) to assess consumers' perceived skills at using information technology for health and (2) to aid in determining the fit between eHealth programs and consumers. Norman, 2006
Health literacy and Ehealth literacy scales (eHEALS) | 18 months
  The eHealth Literacy Scale measures (1) to assess consumers' perceived skills at using information technology for health and (2) to aid in determining the fit between eHealth programs and consumers. Norman, 2006
Health literacy and Ehealth literacy scales (eHEALS) | 24 months
  The eHealth Literacy Scale measures (1) to assess consumers' perceived skills at using information technology for health and (2) to aid in determining the fit between eHealth programs and consumers. Norman, 2006
Health related status | baseline
  Questions include: smoking status, falls, serious health events
Health related status | 6 months
  Questions include: smoking status, falls, serious health events
Health related status | 12 months
  Questions include: smoking status, falls, serious health events
Health related status | 18 months
  Questions include: smoking status, falls, serious health events
Health related status | 24 months
  Questions include: smoking status, falls, serious health events
PROMIS Cognitive Function + PROMIS Cognitive Abilities - 8a | baseline
  Developed, evaluated, and distributed by the National Institutes of Health to measure perceived cognitive functioning
PROMIS Cognitive Function + PROMIS Cognitive Abilities - 8a | 6 months
  Developed, evaluated, and distributed by the National Institutes of Health to measure perceived cognitive functioning
PROMIS Cognitive Function + PROMIS Cognitive Abilities - 8a | 12 months
  Developed, evaluated, and distributed by the National Institutes of Health to measure perceived cognitive functioning
PROMIS Cognitive Function + PROMIS Cognitive Abilities - 8a | 18 months
  Developed, evaluated, and distributed by the National Institutes of Health to measure perceived cognitive functioning
PROMIS Cognitive Function + PROMIS Cognitive Abilities - 8a | 24 months
  Developed, evaluated, and distributed by the National Institutes of Health to measure perceived cognitive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
We agree to share any remaining biospecimens, including plasma, sera, and buffy coat (some stored in RNAlater® and some stored alone). Samples will be accompanied by a limited dataset of deidentified participant data that investigators need for analyses. To facilitate the data sharing, we plan to build a central archive that will allow public access to data dictionaries and limited-access anonymized datasets. We will develop a single password protected Share Point web system so that all data dictionaries, documentation, and data accessibility will have a consistent user interface. All datasets will conform to the "Standards for Privacy of Individually Identifiable Health Information" rule of the Health Insurance Portability and Accountability Act (HIPAA). Data will be made available as either a SAS export dataset, or as a tab-delimited ASCII file.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data and samples will be made available to outside investigators after all aims of the P01 and all primary outcomes papers have been published (consonant with the NIH definition of "timely fashion." Requests for data or biologic samples will be handled on a case-by-case basis, and in consultation with the P01 principal investigators (Dr. Demark-Wahnefried) and other members of the investigative team.
Access Criteria: Requests for data or biologic samples will be handled on a case-by-case basis, and in consultation with the P01 principal investigators (Dr. Demark-Wahnefried) and other members of the investigative team. Individuals in receipt of data and samples must produce proof of human subjects and HIPAA training. For the transfer of biospecimens, Human Materials and Data Transfer Agreements will be established between UAB and the requesting institution. Publications resulting from the transfer of samples or data must credit the P01 grant. For data only, requesting users will be required to sign a data-use sharing agreement.

REFERENCES:
- [Background] Pekmezi D, Fontaine K, Rogers LQ, Pisu M, Martin MY, Schoenberger-Godwin YM, Oster RA, Kenzik K, Ivankova NV, Demark-Wahnefried W. Adapting MultiPLe behavior Interventions that eFfectively Improve (AMPLIFI) cancer survivor health: program project protocols for remote lifestyle intervention and assessment in 3 inter-related randomized controlled trials among survivors of obesity-related cancers. BMC Cancer. 2022 Apr 29;22(1):471. doi: 10.1186/s12885-022-09519-y. PMID 35488238
- [Result] Ivankova NV, Rogers LQ, Herbey II, Martin MY, Pisu M, Pekmezi D, Thompson L, Schoenberger-Godwin YM, Oster RA, Fontaine K, Anderson JL, Kenzik K, Farrell D, Demark-Wahnefried W. Features That Middle-aged and Older Cancer Survivors Want in Web-Based Healthy Lifestyle Interventions: Qualitative Descriptive Study. JMIR Cancer. 2021 Oct 6;7(4):e26226. doi: 10.2196/26226. PMID 34612832
- [Result] Pisu M, Omairi I, Hoenemeyer T, Halilova KI, Schoenberger YM, Rogers LQ, Kenzik KM, Oster RA, Ivankova NV, Pekmezi D, Fontaine K, Demark-Wahnefried W, Martin MY. Developing a virtual assessment protocol for the AMPLIFI Randomized Controlled Trial due to COVID-19: From assessing participants' preference to preparing the team. Contemp Clin Trials. 2021 Dec;111:106604. doi: 10.1016/j.cct.2021.106604. Epub 2021 Oct 29. PMID 34757221
- [Result] Rogers LQ, Pekmezi D, Schoenberger-Godwin YM, Fontaine KR, Ivankova NV, Kinsey AW, Hoenemeyer T, Martin MY, Pisu M, Farrell D, Wall J, Waugaman K, Oster RA, Kenzik K, Winters-Stone K, Demark-Wahnefried W. Using the TIDieR checklist to describe development and integration of a web-based intervention promoting healthy eating and regular exercise among older cancer survivors. Digit Health. 2023 Jun 26;9:20552076231182805. doi: 10.1177/20552076231182805. eCollection 2023 Jan-Dec. PMID 37434730
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688
- See also: Website for those interested in joining the study. — http://amplifymyhealth.org